CLINICAL TRIAL: NCT02432157
Title: Hypertonic Saline Solution in Aneurysmal Subarachnoid Hemorrhage: A Randomized - Phase II Single Blinded Clinical Trial
Brief Title: Safety and Feasibility of Hypertonic Saline Solution After Aneurysmal Subarachnoid Hemorrhage:
Acronym: HS3
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Thomas Jefferson University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 14D.557
Record Dates: First submitted 2015-03-10; First posted 2015-05-04 (Estimated); Last update posted 2016-02-11 (Estimated); Status verified 2016-02

CONDITIONS: Subarachnoid Hemorrhage; Cerebral Vasospasm; Hyponatremia
MeSH Terms: conditions — Subarachnoid Hemorrhage; Vasospasm, Intracranial; Hyponatremia | interventions — 5-(3-hydroxybenzoyl)-2-thiophenesulfonamide

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Hypertonic saline (HTS) (Experimental): A protocol of prophylactic 3% HTS as a volume expander with bolus (over 30 minutes) of 3% HTS at a dose of 250 ml every 6 hours for 7 days. This will be given through a central line as soon as possible and within 72 hours of onset of SAH symptoms.
  Interventions: Drug: HTS 3%
- Standard fluid (Active Comparator): Routine fluid management strategy as pre-specified by our SAH management protocol at Jefferson University Hospital according to the American Heart Association and Neurocritical Care Guidelines for the management of SAH (this includes conventional intravenous fluids or normal saline solutions to maintain a normal hydration status and guided by the treating doctor and daily assessments of fluid balance).
  Interventions: Drug: Standard fluid management

INTERVENTIONS:
Drug: HTS 3% — 3% HTS at a dose of 250 ml every 6 hours for 7 days
  Arms: Hypertonic saline (HTS)
Drug: Standard fluid management — Routine fluid management strategy as pre-specified by our SAH management protocol.
  Arms: Standard fluid

SUMMARY:
Subarachnoid hemorrhage (SAH) occurs after rupture of cerebral aneurysms. Treatment of SAH focuses on avoiding medical complications including cerebral vasospasm, which may result in limited circulation to the brain. Cerebral vasospasm, or thinning of the arteries of the brain, is a feared complication that could potentially cause stroke and worst outcomes after SAH. Hypertonic saline (HTS) is a compound that may be used to prevent vasospasm following SAH by enhancing the circulation in the brain. This study will evaluate if a protocol of volume expansion with HTS is safe and effective in patients with subarachnoid hemorrhage for the prevention of cerebral vasospasm.

DETAILED DESCRIPTION:
This is a prospective, single-center, interventional, randomized, parallel, two-arm (1:1) phase II clinical trial with blinded end-point ascertainment designed to determine the safety and feasibility of a protocol of 3% hypertonic saline (HTS) as a "volume expander" administered within 72-hours of admission and up to 7-days in SAH patients compared to standard fluid management, in individuals with aneurysmal SAH. A common sequela of aneurysmal SAH is vasospasm, which causes significant morbidity and mortality. In addition, 30% of patients with SAH develop hypovolemic hyponatremia (serum sodium [Na] <130mEq/L), predisposing them to develop cerebral ischemia. Current guidelines for the management of aneurysmal SAH recommend: (1) maintaining euvolemia in order to prevent delayed cerebral ischemia (DCI) and (2) using HTS as a treatment option for the prevention and treatment of hypovolemic hyponatremia. Treatment for vasospasm includes induction of hypertension, along with systemic and/or intra-arterial administration of calcium channel blockers, or angioplasty. The investigators will (1) measure the incidence of severe adverse events from our protocol of HTS, (2) measure the incidence of cerebral vasospasm in patients treated with our protocol of HTS as compared to patients treated with standard fluid therapy; and (3) assess the burden of hypovolemic hyponatremia.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 to 70 inclusive
2. Hunt-Hess score of 1-5
3. Glascow Come Scale 4-15
4. Modified Fisher Grade 1-4
5. At least one reactive pupil
6. A brain CT/ MRI demonstrating SAH
7. DSA (digital subtraction angiogram) or CTA confirmed presence of intracranial aneurysm
8. The patient can be started on HTS within 72 hours of onset of symptoms of SAH
9. Previously placed central line or having other indication for central line placement

Exclusion Criteria:

1. Pregnancy, or inability to rule out pregnancy with a pregnancy test
2. A normal head CT scan or a CT scan showing a bleed that is not SAH
3. Spinal cord injury or other serious noncerebral injury
4. Known seizure disorder
5. Known brain disease (eg tumor, metastasis) or major psychiatric disorders (eg schizophrenia)
6. Renal insufficiency (baseline Cr>1.5 mg/dl, CrCl<30 ml/min, CKD)
7. Acute systolic dysfunction or congestive heart failure (CHF), with EF <30%
8. Hematologic abnormalities or coagulopathy (PT>20, PTT>50, INR>1.5, or bleeding time>10sec)
9. Clinically significant cardiovascular, hepatic or pulmonary disease that, in the opinion of the investigator, would compromise patient safety
10. Other life-threatening injury that compromises patient survival through duration of study
11. Patient unlikely to be available for follow-up at 6 months after trial conclusion
12. Any concurrent relevant condition that makes the patient unsuitable for participation or follow-up
13. Serum sodium > 155 mEq/L

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2015-01; Primary Completion 2017-01 (Estimated)

PRIMARY OUTCOMES:
Safety (adverse events) | 21 days
  Incidence or proportion of serious adverse events
Feasibility (Proportion of patients treated according to the protocol) | 21 days
  Proportion of patients treated according to the protocol

SECONDARY OUTCOMES:
Vasospasm (Incidence of cerebral vasospasm defined as clinical deterioration) | 21 days
  Incidence of cerebral vasospasm defined as clinical deterioration (focal deficit or decline in Glasgow Coma Scale (GCS) score of >/=2 points by neurological exam), or transcranial doppler (TCD) velocity increase with mean blood flow > 120 cm/sec, or arterial narrowing (mod-sec) on DSA or CTA.
Hyponatremia (Incidence of hypovolemic hyponatremia defined as Na <135) | 21 days
  Incidence of hypovolemic hyponatremia defined as Na <135

CONTACTS AND LOCATIONS:
Locations (1):
- Thomas Jefferson University Hospital, Philadelphia, Pennsylvania, United States